CLINICAL TRIAL: NCT02162628
Title: Exair® Prolapse Repair System Versus Native Tissue Repair for Treatment of Pelvic Organ Prolapse, Exair 522 Study
Brief Title: Exair® Versus Native Tissue Repair for Prolapse
Status: Terminated | Type: Observational
Why Stopped: Device voluntarily withdrawn from commercial use by manufacturer
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: SU019
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Floor Disorder; Pelvic Organ Prolapse; Sexual Dysfunction; Mesh; POP; Transvaginal; Total Repair; Uterine Prolapse; Cystocele; Rectocele; Enterocele; Vaginal Vault Prolapse; Native Tissue Repair; Repair Augmented with Mesh; Pathological Conditions, Anatomical; Exair Prolapse Repair System; Vaginal Mesh; Transvaginal Mesh
MeSH Terms: conditions — Pelvic Organ Prolapse; Pelvic Floor Disorders; Sexual Dysfunction, Physiological; Uterine Prolapse; Cystocele; Rectocele; Hernia; Pathological Conditions, Anatomical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exair for Total Repair: Total repair with Exair Prolapse Repair System alone or in combination with native tissue repair
  Interventions: Device: Exair Prolapse Repair System
- Total Native Tissue Repair: Total repair with native tissue only
  Interventions: Procedure: Total Native Tissue Repair

INTERVENTIONS:
Device: Exair Prolapse Repair System
  Groups: Exair for Total Repair
Procedure: Total Native Tissue Repair
  Groups: Total Native Tissue Repair

SUMMARY:
The purpose of this study is to compare safety and effectiveness of the Exair Prolapse Repair System for treatment of pelvic organ prolapse to traditional native tissue repair through 36 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female at least 18 years of age
* Subject has pelvic organ prolapse with leading edge at or beyond the hymen. At or beyond the hymen is defined as POP-Q scores of Ba ≥0 and Bp ≥0 and C≥ -1/2 tvl
* Subject reports a bothersome bulge they can see or feel per PFDI-20 question 3, response of 2 or higher (i.e. responses of "somewhat", "moderately" or "quite a bit")
* Subject is willing to provide written informed consent
* Subject is willing and able to comply with the follow-up regimen

Exclusion Criteria:

* Subject is pregnant or intends to become pregnant during the study
* Subject has an active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI), or tissue necrosis
* Subject has a history of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical)
* Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area
* Subject has taken systemic steroids (within the last month), or immunosuppressive or immunomodulatory treatment (within the last 3 months)
* Subject has a systemic connective tissue disease (e.g. scleroderma, systemic lupus erythematosus (SLE), Marfan syndrome, Ehlers Danlos, collagenosis, polymyositis or polymyalgia rheumatica)
* Subject has chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis
* Subject has uncontrolled diabetes mellitus (DM)
* Subject has a known neurologic or medical condition affecting bladder function (e.g. multiple sclerosis, spinal cord injury, or stroke with residual neurologic deficit)
* Subject is seeking obliterative vaginal surgery as treatment for pelvic organ prolapse (colpocleisis)
* Subject is not able to conform to the modified dorsal lithotomy position
* Subject is currently participating in or plans to participate in another device or drug study during this study
* Subject has a known sensitivity to polypropylene
* Subject has had previous prolapse repair with mesh in the target compartment(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with pelvic organ prolapse who are candidates for transvaginal surgical repair.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of Prolapse | 36 Month
  Recurrent prolapse is measured anatomically at the target compartment by leading edge of prolapse beyond the hymenal ring by POP-Q examination, or additional surgical treatment for pelvic organ prolapse in the target vaginal compartment(s), or patient reporting symptoms of vaginal bulging.
Rate of device and procedure related adverse events | 36 Month

SECONDARY OUTCOMES:
Recurrence of prolapse | 36 Month
  Recurrent prolapse is measured anatomically by leading edge of prolapse in the target compartment at or beyond the hymenal ring by POP-Q examination, or additional surgical treatment for pelvic organ prolapse in the target vaginal compartment(s), or patient reporting symptoms of vaginal bulging.
Rates of other adverse events | 36 months

OTHER OUTCOMES:
Changes in Quality of Life scores for PFDI-20, PISQ-12, and PFIQ-7 | 36 months
Subjects experiencing vaginal bulge | 36 months
Rates of revision and/or re-surgery | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: James Lukban, DO, FACOG, Principal Investigator — The Pelvic Solutions Center
Locations (14):
- United States (13):
  - Progressive GYN Center, Savannah, Georgia
  - Women's Health Advantage, Fort Wayne, Indiana
  - Advanced Urogynecology of Michigan, Dearborn, Michigan
  - Minnesota Women's Care, Maplewood, Minnesota
  - Atlantic Urogynecology Associates, Morristown, New Jersey
  - Princeton Urogynecology, Princeton, New Jersey
  - Albany Medical Center, Albany, New York
  - United Health Services, Johnson City, New York
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Novant Health Clinical Research, Winston-Salem, North Carolina
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Vermont Urogynecology Associates, P.C., Williston, Vermont
  - Carillion Clinic OB/GYN, Christiansburg, Virginia
- CHUS-CRC, Sherbrooke, Quebec, Canada